CLINICAL TRIAL: NCT04650503
Title: Clinical Outcome of Mild to Very-mild Asthma With High Sputum Eosinophils and/or High Genetic Risk Score: a Prospective Longitudinal Study
Brief Title: Follow-up of Mild Eosinophilic Asthma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Laval University (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: CÉR21799
Record Dates: First submitted 2020-10-14; First posted 2020-12-02 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-12

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with eosinophilic asthma at baseline: Patients showing ≥3% sputum eosinophils at baseline
  Interventions: Other: No intervention
- Patients with non eosinophilic asthma at baseline: Patients showing <3% sputum eosinophils at baseline
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Asthma is a chronic respiratory disease affecting approximately 10% of the population, the majority of patients with very mild to mild asthma. Asthma is characterized primarily by the presence of symptoms clinical variables, reversible airway obstruction and airway hyperresponsiveness. Inflammation is a key factor in the pathophysiology of the disease. Eosinophilic inflammation is the most common type. However, in the literature it is usually associated with more severe and difficult to control asthma. Although mortality associated with asthma has drastically decreased in recent years, several events still occur. Strangely enough, these frequently affect mild asthmatics. Although there is still a misunderstanding in relation to these events, the most recent practice guides have recommended an approach based on the use of inhaled corticosteroids (ICS) in all, including mild asthmatics. This change of therapeutic cap is still debated, but indicates a need for new studies in this population. Recently, the investigators demonstrated that a subgroup of asthma patients with mild asthma had a eosinophilia. The evolution of this subgroup without bronchial obstruction or respiratory symptoms remains unknown. Indeed, it seems imperative to determine the fate of these subjects in comparison with asthma mild non-eosinophilic since it could be a subgroup at risk of poor outcome. The objective of this study will be to examine the course of asthma in very mild to mild asthma patients who exhibit eosinophilic inflammation of the respiratory tract compared to noneosinophilic subjects.

This will be a prospective observational, longitudinal study. Participants for whom a result of induced sputum showing an eosinophil level greater than or equal to 3% was observed at least 1 year ago will be contacted to participate in the study. They will be matched for age, gender and duration of asthma to subjects without eosinophilia. These subjects will not be on bronchial anti-inflammatory medication. They will have a complete evaluation including respiratory function tests, a methacholine challenge and sputum induction. They will also complete questionnaires on controlling their asthma and exacerbations.

ELIGIBILITY:
Inclusion Criteria:

* With a proven diagnosis of asthma
* With very mild or mild asthma at the time of previous assessment
* With at least two sputum cell differential counts > 1 year before follow-up visit
* With stable asthma and asthma medication for at least 4 weeks before baseline assessment and before follow-up visit
* Able and willing to consent to study procedures

Exclusion Criteria:

* Conditions that could affect measurements, such as any active chronic or systemic inflammatory disease, not related to the respiratory system.
* Subjects with a main diagnosis of eosinophilic granulomatosis with polyangiitis (Churg- Strauss syndrome) or hypereosinophilic syndrome.
* Respiratory tract infection in the 4 weeks preceding past assessments and in the 4 weeks preceding follow-up visit.
* Asthma exacerbation in the 4 weeks preceding past assessments in the 4 weeks preceding follow-up visit.
* Current smokers. Ex-smokers must not have smoked for a minimum of 12 months, and should not have a smoking history ≥10 pack years. Subjects who administer nicotine in other forms (patches, chew tobacco, electronic cigarettes, etc.) will also be excluded from the study;
* Concomitant disease or condition which could interfere with the conduct of the study, or for which the treatment might interfere with the conduct of the study, or which would, in the opinion of the investigator, pose an unacceptable risk to the subject in this study, including, but not limited to, cancer, alcoholism, drug dependency or abuse, or psychiatric disease.
* Pregnant or lactating women at the time of follow-up visit.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asthmatic subjects with at least two sputum cell differential results > 1 year before follow-up visit
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Mean annual change in pre bronchodilator forced expiratory volume in one second (FEV1) and FEV1/forced vital capacity (FVC) between baseline and follow-up between the two groups | At least one year post baseline
  calculated using: (initial value - follow-up value)/number of years between the two tests

SECONDARY OUTCOMES:
Clinical sub score of the Asthma Control Scoring system (ACSS) at follow-up between the two groups | At least one year post baseline
  Score between 20% and 100%
Number of asthma exacerbations in the year preceding follow-up visit between the two groups | At least one year post baseline
  Asthma exacerbations defined as a) number of emergency room visits, b) number of hospitalisations, c) number of oral corticosteroid treatments, and d) number of unscheduled medical visits
Airway reactivity at follow-up between the two groups | At least one year post baseline
  Airway reactivity recorded as methacholine provocative concentration inducing a 20% fall in forced expiratory volume in one second (FEV1) (PC20)
Prescribed therapy at follow-up between the two groups | At least one year post baseline
  Defined as a) daily dose of inhaled corticosteroids (ICS), b) use of second controller therapy
Airway inflammation between the two groups at follow-up | At least one year post baseline
  Percentage of sputum eosinophils
Systemic inflammation between the two groups at follow-up | At least one year post baseline
  Blood levels of eosinophils (X10^9/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Louis-Philippe Boulet, MD, Principal Investigator — IUCPQ-UL
Locations (1):
- Louis-Philippe Boulet, Québec, Canada